CLINICAL TRIAL: NCT06714253
Title: A Phase I/IIa, Dose Escalation Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of Intraductal Administration of RXRG001 to Parotid Gland(s) in Adults With Radiation-Induced Xerostomia and Hyposalivation
Brief Title: Study of Circular RNA Treatment in Patients With Radiation Induced Xerostomia-1
Acronym: SPRINX-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RiboX Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RX-RIX-CS101
Record Dates: First submitted 2024-10-14; First posted 2024-12-03 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Radiation-Induced Xerostomia and Hyposalivation
Keywords: Radiation Induced Xerostomia; First-in-human; Hyposalivation; Circular ribonucleic acid; Aquaporin 1
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: Part 1 (Phase 1): single-arm, open-label Part 2 (Phase 2): randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Investigator
Masking Description: Part 1 (Phase 1): single-arm open-label Part 2 (Phase2): randomized, double-blind, placebo-controlled, parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RXRG001 Part 1 (Experimental): Open-label, single arm with 6 subsequent dose cohorts (3 single dose and 3 multiple dose cohorts) of RXRG001 administered intraductally in the salivary gland (unilateral)
  Interventions: Biological: RXRG001
- RXRG001 Part 2 (Experimental): Randomized double-blind with 3 subsequent multiple dose cohorts. RXRG001 is administered intraductally in the salivary gland (bilateral)
  Interventions: Biological: RXRG001
- Placebo Part 2 (Placebo Comparator): Randomized double-blind with 3 subsequent multiple dose cohorts. Placebo is administered intraductally in the salivary gland (bilateral)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RXRG001 — Circular ribonucleic acid encoding human aquaporin 1 encapsulated in a lipid nanoparticle
  Arms: RXRG001 Part 1; RXRG001 Part 2
Biological: Placebo — Placebo (saline)
  Arms: Placebo Part 2

SUMMARY:
This is a first-in-human clinical study to evaluate the safety, tolerability and efficacy of RXRG001 administered in the ducts of the parotid glands in adult patients with radiation-induced xerostomia (dry mouth) and hyposalivation (reduced saliva production).

In Part 1 of the study (open-label, single-arm), patients will receive unilateral administrations of RXRG001 in 3 single ascending dose cohorts and in 3 multiple ascending dose cohorts.

Part 2 of the study has a randomized, double-blind, placebo-controlled design. Patients will receive bilateral administrations of RXRG001 in 3 multiple ascending dose cohorts.

ELIGIBILITY:
Inclusion Criteria*

1. At least 18 years of age
2. History of radiation treatment or chemoradiotherapy for head and neck cancer for stage 2 or higher
3. Free from recurrence of your cancer and never have had another form of cancer for at least 2 years
4. Suffering from xerostomia and/or hyposalivation and have xerostomia symptoms which were not resolved after treatment for at least 3 months
5. Both parotid glands on imaging examination

Exclusion Criteria*

1. Any active infection
2. Heart failure, reduced kidney function or uncontrolled diabetes (Hemoglobin A1c >=8%)
3. History of autoimmune diseases known to potentially affect the salivary glands
4. Any malignancy, other than head and neck cancer within the past 3 years except for certain skin and cervical cancers
5. Active smoker or use tobacco products or have a history of substance or alcohol abuse

   * Other criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | Part 1: up to 36 weeks, Part 2: up to 36 weeks
  Incidence of treatment-emergent adverse events
Incidence of treatment-emergent serious adverse events | Part 1: up to 36 weeks, Part 2: up to 36 weeks
  Incidence of treatment-emergent serious adverse events

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - John Hopkins University, Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - NYU Langone Medical Center, New York, New York
  - Penn Medicine - Otorhinolaryngology - Head and Neck Surgery Perelman, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No